CLINICAL TRIAL: NCT00006047
Title: Phase I Study of Combination Therapy With Oral 9-Nitrocamptothecin and Oral Etoposide
Brief Title: Combination Therapy With Oral 9-Nitrocamptothecin & Oral Etoposide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-12177; NCI-G00-1821 (Other: NCI)
Record Dates: First submitted 2000-07-05; First posted 2004-02-12 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Etoposide; rubitecan; Topoisomerase I Inhibitors; tocophersolan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination Therapy (Experimental): Combination Therapy with Oral 9-Nitrocamptothecin & Oral Etoposide. Patients receive oral nitrocamptothecin on days 1-3 and oral etoposide on days 4-5 each week. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Oral Etoposide; Drug: Oral 9-Nitrocamptothecin

INTERVENTIONS:
Drug: Oral Etoposide
  Other Names: Vepesid; Oral VP-16
Drug: Oral 9-Nitrocamptothecin
  Other Names: rubitecan; 9NC; oral topoisomerase I inhibitor; PEG-1000

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of nitrocamptothecin plus etoposide in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose, dose limiting toxicity, and safety of nitrocamptothecin when administered with etoposide in patients with advanced solid tumors. II. Determine the changes in expression and activity of topoisomerase I and II which occur during administration of this treatment regimen in these patients. III. Determine the plasma pharmacokinetics of this treatment regimen in these patients. IV. Compare the hematologic and nonhematologic toxicities with this treatment regimen in patients 70 years of age and older versus patients younger than 70 years of age.

OUTLINE: This is a dose escalation study of nitrocamptothecin. Patients receive oral nitrocamptothecin on days 1-3 and oral etoposide on days 4-5 each week. Treatment continues in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of nitrocamptothecin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities. Patients are followed every 4 weeks until toxicities resolve.

PROJECTED ACCRUAL: Approximately 40-60 patients will be accrued for this study over 18 to 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed nonhematologic malignancy refractory to available therapies or for which no curative therapy exists Measurable or evaluable disease No active brain metastases, including evidence of cerebral edema by CT scan or MRI, progression from a prior imaging study, or any requirement for steroids or clinical symptoms of/from brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL ALT and AST less than 2 times upper limit of normal (ULN) (unless clearly related to hepatic metastases) Renal: Creatinine less than 1.5 times ULN Other: No other serious uncontrolled medical disorder or active infection that would preclude study No dementia or altered mental status that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 10 weeks after study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy No concurrent colony stimulating factors (e.g., filgrastim (G-CSF) or sargramostim (GM-CSF)) Chemotherapy: No prior topoisomerase I inhibitors (e.g., nitrocamptothecin, aminocamptothecin, irinotecan, or topotecan) At least 4 weeks since prior chemotherapy (at least 6 weeks since prior nitrosoureas, mitomycin, or carboplatin) No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics At least 4 weeks since prior hormonal therapy No concurrent hormonal anticancer therapy Radiotherapy: At least 4 weeks since prior radiotherapy involving at least 30% of the bone marrow No concurrent radiotherapy Surgery: Not specified Other: No other concurrent experimental anticancer medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2000-06; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 3 years
  Determine the MTD of nitrocamptothecin. Cohorts of 3-6 patients receive escalating doses of nitrocamptothecin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Sullivan, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States